CLINICAL TRIAL: NCT00435201
Title: Characterization of Clonal B Cell Populations in HCV Infection
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Collaborators: New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ECH-0596
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — white blood cells
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the mechanism of autoantibody production during chronic hepatitis C virus (HCV) infection. 10-50% of individuals with HCV have symptoms of mixed cryoglobulinemia (MC). By studying the B cells from HCV-infected individuals with and without MC, as well as from healthy controls, we hope to gain insight into the mechanisms of autoantibody production and develop new strategies for treatment of MC.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infects approximately 170 million people worldwide. About 10-50% of persons with HCV have MC. MC is associated with the development of autoimmune symptoms and B cell proliferative disorders. We plan to study B cells from individuals chronically infected with HCV as well as from healthy controls. We sort B cells into different types, and we analyze these types for differential levels of gene expression. We are testing the hypothesis that certain types of B cells from subjects with MC have increased expression of genes that allow for increased cell survival.

People interested in participating in this study will have a complete history and general medical examinations before beginning the study. Following the screening, you will have a procedure called leukapheresis, in which white blood cells are removed, but your own red blood cells are returned. The procedure takes approximately 3 hours and is similar to blood donation. The leukapheresis is done during a same day admission to the hospital by an outside blood collection company with trained nurses and certified equipment.

Some aspects of this study are experimental which means the fluid and cells collected will be studied and analyzed to determine more precisely how your body's immune system is responding to the virus. These tests are experimental in that they are not part of the usual routine care of patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Ability to give informed consent.
* WBC greater than 3,000/mm3.
* Platelets greater than 80,000/mm3.
* Hb at least 9.5 g/dl.
* INR less than 1.5.
* Biologic therapy: Greater than 6 months post-Rituximab therapy.
* Greater than 6 months post IFN- alpha and Ribavirin therapy.

Exclusion Criteria:

* Decompensated cirrhosis.
* Serious uncontrolled medical illness.
* Receipt of immune modulators or suppressors within 30 days prior to study entry, including, but not limited to, interferons and thalidomide.
* Psychiatric illness or social condition that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Alcohol or drug use or dependence that, in the opinion of the investigator,would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NYC area
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2007-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Dustin, PhD, Principal Investigator — Rockefeller University
Locations (2):
- Rockefeller University Hospital, New York, New York, United States
- Oxford University, Oxford, United Kingdom

REFERENCES:
- [Derived] Charles ED, Brunetti C, Marukian S, Ritola KD, Talal AH, Marks K, Jacobson IM, Rice CM, Dustin LB. Clonal B cells in patients with hepatitis C virus-associated mixed cryoglobulinemia contain an expanded anergic CD21low B-cell subset. Blood. 2011 May 19;117(20):5425-37. doi: 10.1182/blood-2010-10-312942. Epub 2011 Mar 18. PMID 21421840
- See also: Related Info — http://www.rucares.org